CLINICAL TRIAL: NCT04009954
Title: Post-operative Ileus of Colorectal Cancer Patients Associated With Perioperative Gut Microbiota
Brief Title: Post-operative Ileus and Gut Microbiota
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Yunwei Wei 2019-04-19
Record Dates: First submitted 2019-05-13; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Post-operative Ileus
Keywords: Post-operative Ileus; Gut Microbiota; perioperative period
MeSH Terms: interventions — Defecation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Fecal sample analysis will consist of the following procedure : Microbial DNA extraction, amplicon library construction, sequencing and analysis; Clustering "MiSeq" reads into operational taxonomic units (OTUs).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delayed transit: CRC patients with delayed gut transit recovery( first time defecation >3 day )
  Interventions: Other: Fecal and blood samples collection for analysis
- Normal transit: CRC patients with normal gut transit recovery( first time defecation <=3 day )
  Interventions: Other: Fecal and blood samples collection for analysis

INTERVENTIONS:
Other: Fecal and blood samples collection for analysis — Fecal sample analysis will consist of the following procedure : Microbial DNA extraction, amplicon library construction, sequencing and analysis; Clustering "MiSeq" reads into operational taxonomic units (OTUs).

SUMMARY:
Postoperative ileus (POI) is a common clinical condition after abdominal surgical procedure, leading to increased patient morbidity and prolonged hospitalisation.The mechanism of POI is not very clear until now. At the end of the 20th century, the inflammatory-mediated ileus hypothesis was introduced. But the initial trigger of the inflammatory cascade is unclear.Previous study demonstrate a clear association between colonic transit time, gut microbiota composition and urinary metabolic phenotype. Here the investigators suggest that the perioperative gut microbiota may contribute to POI.

DETAILED DESCRIPTION:
Postoperative ileus (POI) is a common clinical condition after abdominal surgical procedure, leading to increased patient morbidity and prolonged hospitalisation.

The clinical manifestations include abdominal distension, nausea, vomiting and the inability to pass stools or tolerate a solid diet. In addition to the discomfort experienced by patients, postoperative ileus is also an important risk factor for complications such as wound dehiscence and pulmonary and thromboembolic complications. Ileus was found to be an important predictor of extended postoperative hospital stays and costs in patients undergoing colectomy.

The mechanism of POI is not very clear until now. At the end of the 20th century, the inflammatory-mediated ileus hypothesis was introduced. But the initial trigger of the inflammatory cascade is unclear The innate immune system recognises two large classes of macromolecules: first, those related to pathogens or pathogen-associated molecular patterns (PAMPs), and secondly, molecules released in response to cell damage or damage-associated molecular patterns (DAMPs). The prototype of PAMPs is lipopolysaccharide (LPS), a constituent of the Gram-negative bacterial cell wall. Translocation of microbial products into the intestinal tissue is a well-documented feature in POI. Previous study demonstrate a clear association between colonic transit time, gut microbiota composition and urinary metabolic phenotype. Here the investigators suggest that the perioperative microbiome may contribute to POI. This study apply NGS(next generation sequencing) technique to analyse the composition of the perioperative gut microbiota of CRC(colorectal cancer) patients, then analysis the relationship between the dynamic variation of gut microbiota and POI.

ELIGIBILITY:
Inclusion Criteria:

* Requirements of informed consent and assent of participant, parent or legal guardian as applicable
* Patients with colorectal cancer scheduled for radical coloproctectomy and between the age of 35 and 80 years old without considering sex.
* Patients with BMI= 18.5-23.9

Exclusion Criteria:

* Patients with colorectal cancer with distant metastasis
* Chronic renal diseases and hepatic cirrhosis
* Chronic ischemic heart disease with unstable angina, chronic heart failure at class III or IV and acute myocardial infarction in the last 6 months
* Individuals with a history of Chronic diarrhea
* Individuals with a history of Diabetes mellitus
* Individuals with a history of Hypertension
* Individuals with a history of autoimmune diseases
* Use of antibiotics and probiotics 3 mouth before samples collection
* Individuals with a history of abdominal operation due to any reason
* Individuals with any history of cancer other than colorectal cancer
* Individuals with Inflammatory bowel disease

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants are patients need undergo an exhaustive colorectal cancer surgical resection in the First Affiliated Hospital of Harbin Medical University from May 1, 2018 to Dec 31, 2019.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in gut microbiome dynamics in colorectal cancer patients during the perioperative period between two groups | The day before operation day, the first to the 10th day after operation (everyday the patient's faeces will be collected for microbiome analysis, if the patient has no faeces,we will skip that day to next day for fecal collection)
  The diversity, structure of fecal microbiota and relative abundance of special bacterial taxa 16S rRNA gene sequencing will be performed.
The time ranging from operation day to the day of first defecation | Up to 10 days
  The recovery of gut transit can be indicated by the first defecation

SECONDARY OUTCOMES:
Concentration of plasma i-FABP(intestinal fatty acid-binding protein) | The day before operation day, every day from first to fifth post-operative day
  The detection of i-FABP is useful to determine localized changes in intestinal damage.
Concentration of plasma LPS | The day before operation day, every day from first to fifth post-operative day
  The presence of lipopolysaccharide (LPS) has been used as an indirect measurement of bacterial translocation and systemic exposure to bacteria.
Concentration of fecal LPS | The day before operation day, the first to the 10th day after operation (everyday the patient's faeces will be collected for microbiome analysis, if the patient has no faeces,we will skip that day to next day for fecal collection)
  LPS was derived from gram-negative bacteria in the intestinal tract, and LPS in blood was derived from feces.
Concentration of fecal calprotectin | The day before operation day, the first to the 10th day after operation (everyday the patient's faeces will be collected for microbiome analysis, if the patient has no faeces,we will skip that day to next day for fecal collection)
  Fecal calprotectin is not only an indicator of intestinal inflammation, but also an indicator of intestinal mucosal barrier.

CONTACTS AND LOCATIONS:
Overall Officials: Yunwei Wei, Study Director — First Affiliated Hospital of Harbin Medical University
Locations (1):
- First affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No